# PVP-Guided Decongestive Therapy in HF 2 (PERIPHERAL-HF2)

NCT06495892

July 1st, 2024

#### Identification

| Project ID# | <br> | _ |
|---|---|---|
| Name and surname | | _ |
| National ID# | | |
| Age | | |
| Gender | nale | - |
| Boy<br>(in centimeters) | | _ |
| Kilo<br>(the first measured weight in kilograms) | | _ |
| Recommend allowing access for physicians to e-pulse account. (For easy access to long-term follow-up). | | |
| Phone number<br>(May be required for follow-up. Example; 0532 510 97<br>98, 0216 283 38 38) | | _ |
| Phone number #2 (if available)<br>(May be required for follow-up. Example; 0532 510 97<br>98, 0216 283 38 38) | | _ |



#### Randomization

| Center (Please select randomizing center.) | <ul> <li>Ankara Etlik Şehir Hastanesi</li> <li>Antalya Atatürk Devlet Hastanesi</li> <li>Akdeniz Üniversitesi Tıp Fakültesi</li> <li>Bağcılar Eğitim ve Araştırma Hastanesi</li> <li>Bakırçay Üniversitesi Tıp Fakültesi, Çiğli Eğitim ve Araştırma Hastanesi</li> <li>Başakşehir Çam ve Sakura Şehir Hastanesi</li> <li>Dr. Siyami Ersek Göğüs Kalp ve Damar Cerrahisi Eğitim Ve Araştırma Hastanesi</li> <li>Eskişehir Şehir Hastanesi</li> <li>Erzurum Atatürk Üniversitesi Hastanesi</li> <li>İdil Devlet Hastanesi</li> <li>Kafkas Üniversitesi Sağlık Araştırma ve Uygulama Hastanesi</li> <li>Kütahya Sağlık Bilimleri Üniversitesi Tıp Fakültesi Hastanesi</li> <li>Mehmet Akif Ersoy Eğitim ve Araştırma Hastanesi</li> <li>Pazarcık Devlet Hastanesi</li> <li>Tokat Gaziosmanpaşa Üniversitesi Tıp Fakültesi Hastanesi</li> <li>Trakya Üniversitesi Tıp Fakültesi Hastanesi</li> </ul> |
|---|---|
| Study arm (Study arm according to randomization scheme) | <ul><li>○ Pressure guided</li><li>○ Standard</li></ul> |
| Randomization date<br>(Select as day-month-year) | |
| Has the patient been excluded? (Has the patient been excluded after randomization ?) | ○ Yes<br>○ No |
| Select the reason for exclusion. (Select the reason for exclusion if the patient has been excluded after randomization.) | <ul> <li>Upper extremity venous disease</li> <li>Serum creatinine ≥ 3.5 mg/dL</li> <li>Severe stenotic valvular disease</li> <li>Hypertrophic obstructive cardiomyopathy</li> <li>Rejection or withdrawal of consent</li> <li>Other</li> </ul> |
| Please explain. (Explain the reason for exclusion if the patient has been excluded after randomization.) | |
| Consent form (You can download consent form from this link.) | |
| [Attachment: "PERIPHERAL-HF Onam formu.pdf"] | |
| Signed consent form | |
| (Please upload scanned file or photo of signed consent form. Keep the original.) | |



#### History

| Project ID# | | |
|---|---|---|
| Hypertension (Average blood pressure >140/90 mmHg or use of antihypertensive medication) | ○ Yes | ○ No |
| Diabetes (FPG>126 mg/dL for two times or HbA1c>%6.5 or use of antidiabetic medication) | ○ Yes | ○ No |
| Dyslipidemia | ○ Yes | ○ No |
| (LDL>160 mg/dL or use of antihyperlipidemic drug) | | |
| Active smoking (Smoking history in the last one year) | ○ Yes | ○ No |
| Chronic obstructive pulmonary disease<br>(Prior diagnosis of COPD or long-acting bronchodilator<br>use with a clinical picture consistent with COPD) | ○ Yes | ○ No |
| Chronic kidney disease<br>(GFR < 60 ml/min/1.73 m2 known or supposed to be<br>longer than 3 months) | ○ Yes | ○ No |
| Prior myocardial infarct<br>(Documented diagnosis or imaging evidence of an old<br>[>1 month] myocardial infarct) | ○ Yes | ○ No |
| Prior percutaneous coronary intervention | ○ Yes | ○ No |
| (Documented history or imaging evidence of a prior coronary intervention) | | |
| Prior coronary arterial by-pass grafting<br>(Documented history or imaging evidence of a prior<br>CABG) | ○ Yes | ○ No |
| Prior ICD/CRT implantation (Documented history or imaging evidence of a prior ICD/CRT implantation) | ○ Yes | ○ No |



#### **Admission Findings**

| Admission type<br>(With regard to heart failure) | <ul><li>De novo heart failure</li><li>Heart failure decompensation</li></ul> |
|---|---|
| Etiology of heart failure<br>(Respond accoerding to current or past information.) | <ul><li>○ Ischemic</li><li>○ Non-ischemic</li><li>○ Could not be differentiated</li></ul> |
| Systolic blood pressure on admission (in mmHg) | |
| Heart rate on admission<br>(in beats per minute) | |
| Subjective dyspnea score | |
| <ul><li>None</li><li>Rare</li><li>Frequent</li><li>Always</li></ul> | |
| Subjective orthopnea score | |
| <ul><li>None</li><li>Rare</li><li>Frequent</li><li>Always</li></ul> | |
| Subjective fatigue score | |
| <ul><li>○ None</li><li>○ Rare</li><li>○ Frequent</li><li>○ Always</li></ul> | |
| Pretibial edema | |
| <ul><li>○ None</li><li>○ 1+</li><li>○ 2+</li><li>○ 3+</li><li>○ 4+</li></ul> | |
| Pulmonary rales | |
| <ul><li>○ None</li><li>○ Limited to the bases</li><li>○ Lower half</li><li>○ More than lower half</li></ul> | |



| Jugular venous distention | |
|---|---|
| (Compared to angle of Louis while lying at 45 degree supine | position.) |
| <ul><li>○ Cannot be observed</li><li>○ Normal (&lt; 4.5 cm)</li><li>○ High (&gt;4.5 cm) but pulsations can be seen</li><li>○ Exceeds angulus mandibula</li></ul> | |
| BUN on admission (Just before or after admission, in mg/dL, e.g.; 12) | |
| Creatinine on admission (Just before or after admission, in mg/dL, e.g.; 1.2) | |
| Sodium on admission<br>(Just before or after admission, in mEq/L, e.g.; 142) | |
| Potassium on admission (Just before or after admission, in mEq/L, e.g.; 4.2) | |
| Hemoglobin on admission (Just before or after admission, in g/dL, e.g.; 12.3) | |
| Hematocrit on admission (Just before or after admission, in %, e.g.; 31) | |
| Albumin on admission (Just before or after admission, in g/dL, e.g.; 3.1) | |
| Total protein on admission (Just before or after admission, in g/dL, e.g.; 5.2) | |
| BNP/NT-proPNP on admission (Just before or after admission, in pg/mL, e.g.; 125) | |
| Uric acid on admission (Just before or after admission, in mg/dL, e.g.; 5.5) | |
| Rhythm on ECG ?<br>(Dominant rhythm on ECG') | <ul><li>○ Sinus</li><li>○ AF</li><li>○ Other</li></ul> |
| Left bundle branch block on ECG ?<br>(Select according to the dominant conduction, excluding pacemaker rhythm) | ○ Yes<br>○ No |
| Ejection fraction<br>(in percent, example; 55) | |
| Mitral regurgitation (0=none, 1=mild, 2=moderate, 3=moderate-to-severe, | |



| Tricuspid regurgitation (0=none, 1=mild, 2=moderate, 3=moderate-to-severe, 4=severe) | |
|---|---|
| Estimated pulmonary arterial pressure (in mmHg including estimated right atrial pressure, e.g.; 50. 0 if cannot be calculated.) | |
| Venous pressure | |
| (in mmHg; e.g., 5. If the subject is in standard therapy arm, caregiver should be blinded to this measurement.) | |
| Quality of waveform | <ul> <li>Good (Clear atrial or respiratory pressure oscillations)</li> </ul> |
| (Interpret the visual quality of waveform) | <ul> <li>Moderate (Less clear pressure oscillations but a stable measurement with an appropriate modified-Valsalva response)</li> <li>Poor (No oscillations, increasing, no appropriate modified-Valsalva response or nonphysiological readings)</li> </ul> |

#### **Prior Medications**

| Aspirin (Used medications before admission) | ○ Yes | ○ No |
|---|---|---|
| P2Y12 inhibitor<br>(Used medications before admission) | ○ Yes | ○ No |
| OAC/NOAC<br>(Used medications before admission) | ○ Yes | ○ No |
| Beta-blocker<br>(Used medications before admission) | ○ Yes | ○ No |
| ACEi/ARB<br>(Used medications before admission) | ○ Yes | ○ No |
| ARNI<br>(Used medications before admission) | ○ Yes | ○ No |
| SGLT2i<br>(Used medications before admission) | ○ Yes | ○ No |
| MRA (Used medications before admission) | ○ Yes | ○ No |
| Loop diuretic<br>(Used medications before admission) | ○ Yes | ○ No |
| Oral furosemide equivalent dose<br>(40 mg furosemide po=20 mg furosemide iv=20 mg<br>torasemide po) | | |
| Digoxin<br>(Used medications before admission) | ○ Yes | ○ No |
| Statin (Used medications before admission) | ○ Yes | ○ No |



# In-hospital Course (1st day)

| 1st day fluid intake |
|---|
| (From admission to next day morning, in mL , e.g.; 1250) |
| 1st day urine output |
| (From admission to next day morning, in mL, e.g.; 1250. Do not add extra losses, such as paracentesis or thoracentesis) |
| BUN after 1st day |
| (First morning value after admission, in mg/dL , e.g.;<br>25) |
| Creatinine after 1st day |
| (First morning value after admission, in $mg/dL$ , e.g.; 1.5) |
| Sodium after 1st day |
| (First morning value after admission, in mEq/L , e.g.;<br>135) |
| Potassium after 1st day |
| (First morning value after admission, in mEq/L , e.g.; $4.5$ ) |
| Total intravenous furosemide equivalent of loop diuretic dose |
| (40 mg furosemide po=20 mg furosemide iv=20 mg torasemide po) |
| Total asetozolamide dose<br>(0 if not used) |
| Total thiazide dose<br>(0 if not used) |
| Total MRA dose<br>(0 if not used) |
| 1st day venous pressure |
| (Value in the first morning after admission, in mmHg, e.g; 25) |



| Quality of waveform | <ul> <li>Good (Clear atrial or respiratory pressure oscillations)</li> </ul> |
|---|---|
| (Interpret the visual quality of waveform) | <ul> <li>Moderate (Less clear pressure oscillations but a stable measurement with an appropriate modified-Valsalva response)</li> <li>Poor (No oscillations, increasing, no appropriate modified-Valsalva response or nonphysiological readings)</li> </ul> |
| You do not need to input any data in this form as the in-hospital follow-up is ended. Please proceed to the next instrument . (If in-hospital follow-up continues, check the previous form "Discharged today (or follow-up is terminated for another reason)? and change the answer to "No".) | ○ Yes<br>○ No |

## In-hospital Course (2nd day)

| 2nd day fluid intake | |
|---|---|
| (From previous to this day morning, in mL , e.g.; 1250) | - |
| 2nd day urine output | |
| (From previous to this day morning, in mL , e.g.; 1250. Do not add extra losses, such as paracentesis or thoracentesis) | - |
| BUN after 2nd day | |
| (First morning value after admission, in mg/dL , e.g.; 25) | - |
| Creatinine after 2nd day | |
| (First morning value after admission, in mg/dL , e.g.; $1.5$ ) | - |
| Sodium after 2nd day | |
| (First morning value after admission, in mEq/L , e.g.; 135) | - |
| Potassium after 2nd day | |
| (First morning value after admission, in mEq/L , e.g.; 4.5) | - |
| Total intravenous furosemide equivalent of loop diuretic dose | |
| (40 mg furosemide po=20 mg furosemide iv=20 mg torasemide po) | - |
| Total asetozolamide dose<br>(0 if not used) | - |
| Total thiazide dose<br>(0 if not used) | - |
| Total MRA dose<br>(0 if not used) | <br>- |
| 2nd day venous pressure | |
| (Value in the second morning after admission, in mmHg, e.g; 25) | - |



| Quality of waveform (Interpret the visual quality of waveform) | <ul> <li>Good (Clear atrial or respiratory pressure oscillations)</li> <li>Moderate (Less clear pressure oscillations but a stable measurement with an appropriate modified-Valsalva response)</li> <li>Poor (No oscillations, increasing, no appropriate modified-Valsalva response or nonphysiological readings)</li> </ul> |
|---|---|
| Discharged today (or follow-up is terminated for another reason) ? | ○ Yes<br>○ No |
| (If "Yes" these values will be accepted as pre-discharge measurements.) | |



## In-hospital Course (3rd day)

| 3rd day fluid intake |
|---|
| (From previous to this day morning, in mL , e.g.; 1250) |
| 3rd day urine output |
| (From previous to this day morning, in mL , e.g.; 1250. Do not add extra losses, such as paracentesis or thoracentesis) |
| BUN after 3rd day |
| (Third morning value after admission, in mg/dL , e.g.; 25) |
| Creatinine after 3rd day |
| (Third morning value after admission, in mg/dL , e.g.; 1.5) |
| Sodium after 3rd day |
| (Third morning value after admission, in mEq/L , e.g.; 135) |
| Potassium after 3rd day |
| (Third morning value after admission, in mEq/L , e.g.; 4.5) |
| Total intravenous furosemide equivalent of loop diuretic dose |
| (40 mg furosemide po=20 mg furosemide iv=20 mg torasemide po) |
| Total asetozolamide dose<br>(0 if not used) |
| Total thiazide dose<br>(0 if not used) |
| Total MRA dose<br>(0 if not used) |
| 3rd day venous pressure |
| (Value in the third morning after admission, in mmHg, e.g.,; 25) |



| Quality of waveform (Interpret the visual quality of waveform) | <ul> <li>Good (Clear atrial or respiratory pressure oscillations)</li> <li>Moderate (Less clear pressure oscillations but a stable measurement with an appropriate modified-Valsalva response)</li> <li>Poor (No oscillations, increasing, no appropriate modified-Valsalva response or nonphysiological readings)</li> </ul> |
|---|---|
| Discharged today (or follow-up is terminated for another reason) ? | ○ Yes<br>○ No |
| (If "Yes" these values will be accepted as pre-discharge measurements.) | |



## In-hospital Course (4th day)

| 4th day fluid intake |
|---|
| (From previous to this day morning, in mL , e.g.; 1250) |
| 4th day urine output |
| (From previous to this day morning, in mL , e.g.; 1250. Do not add extra losses, such as paracentesis or thoracentesis) |
| BUN after 4th day |
| (Fourth morning value after admission, in mg/dL, e.g.; 25) |
| Creatinine after 4th day |
| (Fourth morning value after admission, in mg/dL , e.g.; 1.5) |
| Sodium after 4th day |
| (Fourth morning value after admission, in mEq/L , e.g.; 135) |
| Potassium after 4th day |
| (Fourth morning value after admission, in mEq/L , e.g.; 4.5) |
| Total intravenous furosemide equivalent of loop diuretic dose |
| (40 mg furosemide po=20 mg furosemide iv=20 mg torasemide po) |
| Total asetozolamide dose<br>(0 if not used) |
| Total thiazide dose<br>(0 if not used) |
| Total MRA dose<br>(0 if not used) |
| 4th day venous pressure |
| (Value in the fourth morning after admission, in mmHg, e.g; 25) |



| Quality of waveform (Interpret the visual quality of waveform) | <ul> <li>Good (Clear atrial or respiratory pressure oscillations)</li> <li>Moderate (Less clear pressure oscillations but a stable measurement with an appropriate modified-Valsalva response)</li> <li>Poor (No oscillations, increasing, no appropriate modified-Valsalva response or nonphysiological readings)</li> </ul> |
|---|---|
| Discharged today (or follow-up is terminated for another reason) ? | ○ Yes<br>○ No |
| (If "Yes" these values will be accepted as pre-discharge measurements.) | |



## In-hospital Course (5th day)

| 5th day fluid intake | |
|---|---|
| (From previous to this day morning, in mL , e.g.; 1250) | |
| 5th day urine output | |
| (From previous to this day morning, in mL, e.g.;<br>1250. Do not add extra losses, such as paracentesis or<br>thoracentesis) | |
| BUN after 5th day | |
| (Fifth morning value after admission, in mg/dL , e.g.;<br>25) | |
| Creatinine after 5th day | |
| (Fifth morning value after admission, in mg/dL , e.g.;<br>1.5) | |
| Sodium after 5th day | |
| (Fifth morning value after admission, in mEq/L , e.g.;<br>135) | |
| Potassium after 5th day | |
| (Fifth morning value after admission, in mEq/L , e.g.;<br>4.5) | |
| Total intravenous furosemide equivalent of loop diuretic dose | |
| (40 mg furosemide po=20 mg furosemide iv=20 mg torasemide po) | - |
| Total asetozolamide dose<br>(0 if not used) | |
| Total thiazide dose<br>(0 if not used) | |
| Total MRA dose<br>(0 if not used) | |
| 5th day venous pressure | |
| (Value in the fifth morning after admission, in mmHg, e.g; 25) | |



| Quality of waveform (Interpret the visual quality of waveform) | <ul> <li>Good (Clear atrial or respiratory pressure oscillations)</li> <li>Moderate (Less clear pressure oscillations but a</li> </ul> |
|---|---|
| (interpret the visual quality of wavelorm) | stable measurement with an appropriate modified-Valsalva response) Poor (No oscillations, increasing, no appropriate modified-Valsalva response or nonphysiological readings) |
| Discharged today (or follow-up is terminated for another reason) ? | <ul><li>○ Yes</li><li>○ No</li></ul> |
| (If "Yes" these values will be accepted as pre-discharge measurements.) | |



## In-hospital Course (6th day)

| 6th day fluid intake | |
|---|---|
| (From previous to this day morning, in mL , e.g.; 1250) | |
| 6th day urine output | |
| (From previous to this day morning, in mL, e.g.;<br>1250. Do not add extra losses, such as paracentesis or<br>thoracentesis) | |
| BUN after 6th day | |
| (Sixth morning value after admission, in mg/dL , e.g.;<br>25) | |
| Creatinine after 6th day | |
| (Sixth morning value after admission, in mg/dL , e.g.; $1.5$ ) | |
| Sodium after 6th day | |
| (Sixth morning value after admission, in mEq/L , e.g.; 135) | |
| Potassium after 6th day | |
| (Sixth morning value after admission, in mEq/L , e.g.; 4.5) | |
| Total intravenous furosemide equivalent of loop diuretic dose | |
| (40 mg furosemide po=20 mg furosemide iv=20 mg torasemide po) | - |
| Total asetozolamide dose<br>(0 if not used) | |
| Total thiazide dose<br>(0 if not used) | |
| Total MRA dose<br>(0 if not used) | |
| 6th day venous pressure | |
| (Value in the sixth morning after admission, in mmHg, e.g; 25) | |



| Quality of waveform (Interpret the visual quality of waveform) | <ul> <li>Good (Clear atrial or respiratory pressure oscillations)</li> <li>Moderate (Less clear pressure oscillations but a stable measurement with an appropriate modified-Valsalva response)</li> <li>Poor (No oscillations, increasing, no appropriate modified-Valsalva response or nonphysiological readings)</li> </ul> |
|---|---|
| Discharged today (or follow-up is terminated for another reason) ? | ○ Yes<br>○ No |
| (If "Yes" these values will be accepted as pre-discharge measurements.) | |



## In-hospital Course (7th day)

| 7th day fluid intake | |
|---|---|
| (From previous to this day morning, in mL , e.g.; 1250) | |
| 7th day urine output | |
| (From previous to this day morning, in mL, e.g.;<br>1250. Do not add extra losses, such as paracentesis or<br>thoracentesis) | |
| BUN after 7th day | |
| (Seventh morning value after admission, in mg/dL , e.g.; 25) | |
| Creatinine after 7th day | |
| (Seventh morning value after admission, in mg/dL , e.g.; $1.5$ ) | |
| Sodium after 7th day | |
| (Seventh morning value after admission, in mEq/L , e.g.; 135) | |
| Potassium after 7th day | |
| (Seventh morning value after admission, in mEq/L , e.g.; 4.5) | |
| Total intravenous furosemide equivalent of loop diuretic dose | |
| (40 mg furosemide po=20 mg furosemide iv=20 mg torasemide po) | - |
| Total asetozolamide dose<br>(0 if not used) | |
| Total thiazide dose<br>(0 if not used) | |
| Total MRA dose<br>(0 if not used) | |
| 7th day venous pressure | |
| (Value in the seventh morning after admission, in mmHg, e.g; 25) | |



| Quality of waveform (Interpret the visual quality of waveform) | <ul> <li>Good (Clear atrial or respiratory pressure oscillations)</li> <li>Moderate (Less clear pressure oscillations but a stable measurement with an appropriate modified-Valsalva response)</li> <li>Poor (No oscillations, increasing, no appropriate modified-Valsalva response or nonphysiological readings)</li> </ul> |
|---|---|
| Discharged today (or follow-up is terminated for another reason) ? | <ul><li>Yes</li><li>No</li></ul> |
| (If "Yes" these values will be accepted as pre-discharge measurements.) | |



#### **In-hospital Adverse Events**

| Technical problems in pressure monitorization | ○ Yes | ○No |
|---|---|---|
| (Unable to measure venous pressure on admission, before pre-discharge or on three consecutive days) | | |
| *Criterion for exclusion from long-term follow-up (If admission and predischarge pressures cannot be measured)! | | |
| Symptomatic hypotension requiring intervention | ○ Yes | ○ No |
| (Systolic blood pressure < 90 mmHg requiring fluid resuscitation or vasopressor use.) | | |
| Any need for high dose inotropes or mechanical support (intraaortic balloon etc.) | ○ Yes | ○ No |
| (>10 mcg/kg/min dopamine or dobutamine, any dose of noradrenaline or adrenaline. Milrinon or levosimendan can be ignored.) | | |
| *Criterion for exclusion from long-term follow-up! | | |
| The development of clinical thrombophylebitis | ○ Yes | ○No |
| (Redness, warmness or tenderness on any previously used vein) | | |
| Any need for veno-venous hemofiltration or dialysis | ○ Yes | ○No |
| (Any unplanned need for veno-venous hemofiltration or dialysis during hospitalization.) | | |
| *Criterion for exclusion from long-term follow-up! | | |
| In-hospital intubation | ○ Yes | ○ No |
| *Criterion for exclusion from long-term follow-up! | | |
| In-hospital cardiopulmonary resuscitation | ○ Yes | ○ No |
| *Criterion for exclusion from long-term follow-up! | | |
| Exclusion date | | |
| In-hospital mortality | ○ Yes | ○ No |
| *Criterion for exclusion from long-term follow-up! | | |
| Mortality date | | |



#### **Predischarge Findings**

As an in-hospital safety endpoint has occured, this patient has been excluded from long-term follow-up. You do not need to fill any measurement on this page. (If this has not occured and you think this is a mistake, please check the form entitled "In-hospital adverse events".) Dischareg date (Select as day, month and year.) Subjective dyspnea score ○ None ○ Rare Frequent ○ Always Subjective orthopnea score None Rare Frequent Always Subjective fatigue score ○ None ○ Rare Frequent Always Pretibial edema ○ None ○ 1+ ○ 2+ **Ŏ** 3+  $\bigcirc$  4+ Pulmonary rales ○ None Limited to the bases O Lower half More than lower half Jugular venous distention (Compared to angle of Louis while lying at 45 degree supine position.) ○ Unobservable ○ Normal (< 4.5 cm)</p> ○ High (>4.5 cm) but pulsations can be seen Exceeds angulus mandibula BUN on discharge (Just before discharge, in mg/dL, e.g.; 12)



| Creatinine on discharge (Just before discharge, in mg/dL, e.g.; 1.2) | |
|---|---|
| Sodium on discharge<br>(Just before or after admission, in mEq/L, e.g.; 142) | <del></del> |
| Potassium on discharge<br>(Just before discharge, in mEq/L, e.g.; 4.2) | |
| Hemoglobin on discharge<br>(Just before discharge, in g/dL, e.g.; 12.3) | |
| Hematocrit on discharge<br>(Just before discharge, in %, e.g.; 31) | |
| Albumin on discharge (Just before discharge, in g/dL, e.g.; 3.1) | |
| Total protein on discharge<br>(Just before discharge, in g/dL, e.g.; 5.2) | |
| BNP/NT-proPNP on discharge (Just before discharge, in pg/mL, e.g.; 125) | |
| Uric acid on discharge<br>(Just before discharge, in mg/dL, e.g.; 5.5) | |
| Weight<br>(Just before discharge, in kilograms) | |
| Additions to total negative balance (Additional fluid losses, such as paracentesis, thoracentesis, in mL. E.g., 1.200. If absent, enter 0.) | |
| Venous pressure | |
| (in mmHg; e.g., 5. If the subject is in standard therapy arm, caregiver should be blinded to this measurement.) | |
| Quality of waveform | <ul> <li>Good (Clear atrial or respiratory pressure oscillations)</li> </ul> |
| (Interpret the visual quality of waveform) | <ul> <li>Oscillations)</li> <li>Moderate (Less clear pressure oscillations but a stable measurement with an appropriate modified-Valsalva response)</li> <li>Poor (No oscillations, increasing, no appropriate modified-Valsalva response or nonphysiological readings)</li> </ul> |



## **Treatment on Discarge**

| As an in-hospital safety endpoint has occured, this patient need to fill any measurement on this page. | has been exclu | ded from long-term follow-up. You do not |
|---|---|---|
| (If this has not occured and you think this is a mistake, please check the form entitled "In-hospital adverse events".) | | |
| Aspirin (Prescribed medications at discharge) | ○ Yes | ○ No |
| P2Y12 inhibitor<br>(Prescribed medications at discharge) | ○ Yes | ○ No |
| OAC/NOAC<br>(Prescribed medications at discharge) | ○ Yes | ○ No |
| Beta-blocker<br>(Prescribed medications at discharge) | ○ Yes | ○ No |
| ACEi/ARB<br>(Prescribed medications at discharge) | ○ Yes | ○ No |
| ARNI<br>(Prescribed medications at discharge) | ○ Yes | ○ No |
| SGLT2i<br>(Prescribed medications at discharge) | ○ Yes | ○ No |
| MRA<br>(Prescribed medications at discharge) | ○ Yes | ○ No |
| Loop diuretic<br>(Prescribed medications at discharge) | ○ Yes | ○ No |
| Oral furosemide equivalent loop diuretic dose (40 mg furosemide po=20 mg furosemide iv=20 mg torasemide po) | | |
| Digoxin<br>(Prescribed medications at discharge) | ○ Yes | ○ No |
| Statin<br>(Prescribed medications at discharge) | ○ Yes | ○ No |



#### Long-term Follow-up

| As an in-hospital safety endpoint has occured, this patient has been excluded from long-term follow-up. You do not need to fill any measurement on this page. | | | |
|---|---|---|---|
| (If this has not occured and you think this is a mistake, please check the form entitled "In-hospital adverse events".) | | | |
| Long-term mortality<br>(Death in the first year) | ○ Yes | ○ No | ○ Unknown |
| Mortality date | | | |
| All-cause long-term hospitalization (Emergency department visit or hospital admission due to any cause in the first year) | ○ Yes | ○ No | ○ Unkonwn |
| Date of all-cause hospitalization<br>(The first date of emergency department visit or<br>hospital admission due to any cause in the first year) | | | |
| Long-term hospitalization due to HF<br>(Emergency department visit or hospital admission due<br>to HF in the first year) | ○ Yes | ○ No | ○ Unknown |
| Date of HF-related hospitalization<br>(The first date of emergency department visit or<br>hospital admission due to HF in the first year) | | | |

